CLINICAL TRIAL: NCT01448382
Title: Evaluation of PillCam With Blood-Sensing Feature: A Feasibility Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RD-401
Record Dates: First submitted 2011-10-04; First posted 2011-10-07 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2015-12

CONDITIONS: Upper GI Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy volunteers (Experimental): healthy volunteers
  Interventions: Device: PillCam® capsule with Given PillCam® Platform
- GI bleeding subjcets (Experimental): Symptomatic patients referred to undergo standard Gastroscopy (EGD) as part of their standard medical care
  Interventions: Device: PillCam® capsule with Given PillCam® Platform

INTERVENTIONS:
Device: PillCam® capsule with Given PillCam® Platform — capsule endoscopy
  Other Names: CE

SUMMARY:
1. Primary Scientific Objective

   * Collect human clinical data to sustain the development of blood detection sensor and optimize its algorithm and parameters
   * Preliminary evaluation of blood detection performances in human.
2. Secondary Scientific Objective

   * Assessment of blood detection sensor ability to identify the anatomical location (i.e. Stomach, SB or Colon)
   * Evaluation of capsule transit characteristics in the GI tract
   * Evaluation of BBC capsule safety

Study Hypothesis:

It is estimated that by implementing a spectrophotometer technology in capsule and utilizing the unique characteristics of light absorption by blood in specific spectrum, the capsule will be able to automatically detect blood in the GI tract with high accuracy. As such, the system may be an add-on to video capsules to provide efficient and quick detection of blood presence (for example in OGBI patients) or as stand alone low cost capsule (without video) which could serve as a tool similar to standard FOBT.

DETAILED DESCRIPTION:
This study is designed to support the development of a novel blood sensing detector embedded in a PillCam® capsule and to provide initial evaluation of its performance in humans. The device is named Blood Sensing Capsule (BSC), and is based on the Given PillCam® Platform with a modified capsule.

ELIGIBILITY:
Inclusion Criteria:

Group A (Healthy subjects)

* Subject's age is 18 to 45 years old
* Subject is an healthy volunteer
* Subject agrees to sign the Informed Consent Form

Group B (Symptomatic Patients)

* Age ≥ 18 years
* The subject was referred to Gastroscopy for at least one of the following reasons:

  1. History of acute, overt UGI hemorrhage, defined as hematemesis (fresh blood or coffee grounds) and/or melena within the 48 hours prior to patient presentation
  2. Subject has ongoing overt gastrointestinal bleeding with hematochezia or melena
  3. Subject has Iron Deficiency Anemia ,FOBT(+) and negative colonoscopy examination
  4. Other known or suspected cause of acute upper GI bleeding
* Subject agrees to sign the Informed Consent Form

Exclusion Criteria:

1. Subject has Dysphagia, odynophagia, known swallowing disorder or history of Zencker's diverticulum
2. Subject is known or is suspected to suffer from bowel obstruction or bowel perforation at the time of presentation
3. Subject has history of prior bowel obstruction
4. Subject suffers UGI hemorrhage with hemodynamic shock requiring urgent endoscopy
5. Subject with any condition believed to have an increased risk for capsule retention such as Crohn's disease, intestinal tumors, radiation enteritis, incomplete colonoscopies due to obstructions or NSAID enteropathy
6. Subject has history of UGI tract surgery (e.g., Billroth I, Billroth II, esophagectomy, gastrectomy, bariatric procedure)
7. Pregnancy or nursing mothers
8. Subject has known allergy to conscious sedation medications
9. Presence of an electro-medical device (pacemaker or internal cardiac defibrillator)
10. Subject has altered mental status (e.g., hepatic encephalopathy) that would limit patient ability in swallowing the capsule
11. Known allergy to erythromycin
12. Subject is currently or within previous 30 days participating in another clinical study that may directly or indirectly affect the results of this study
13. Subject is not able to provide written informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2011-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Agreement level between the blood detectors head to capsule video head in detecting subjects with blood in the GI tract | 1 year

SECONDARY OUTCOMES:
Agreement level between the blood detectors head to capsule video head in detecting subjects with blood per anatomical location (i.e. stomach, small bowel or colon) | 1 year
Number, type and severity of adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Chowers, PhD., Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam medical center, Haifa, Israel